CLINICAL TRIAL: NCT02335905
Title: Phase 1/2 Trial of Ceftaroline for the Treatment of Hematogenously Acquired Staphylococcus Aureus Osteomyelitis in Children
Brief Title: Ceftaroline for Treatment of Hematogenously Acquired Staphylococcus Aureus Osteomyelitis in Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Sheldon Kaplan, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-35130; TEF-IT-43/IIT-2017-10048 (Other Grant/Funding Number: Allergan)
Record Dates: First submitted 2014-12-31; First posted 2015-01-12 (Estimated); Results first posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Hematogenously Acquired Staphylococcus Aureus Osteomyelitis; Bone Infection; Osteomyelitis
MeSH Terms: conditions — Osteomyelitis | interventions — Ceftaroline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ceftaroline Fosamil (Experimental): IV Ceftaroline fosamil 15 mg/kg (or 600 mg if > 40 kg) infused over 120 (± 10) minutes q8h (± 1 hour). The dose may vary with age.
  Interventions: Drug: Ceftaroline Fosamil

INTERVENTIONS:
Drug: Ceftaroline Fosamil — IV Ceftaroline fosamil 15 mg/kg (or 600 mg if > 40 kg) infused over 120 (± 10) minutes q8h (± 1 hour) for children 2 years of age - 17 years of age (inclusive). IV Ceftarloine Fosamil 10 mg/kg infused 120 (± 10) minutes q8h (± 1 hour) for children 1 years of age - less than 2 years of age (inclusive).

SUMMARY:
This research study is looking at an antibiotic medicine, Ceftaroline Fosamil (Ceftaroline), which fights infections like the one the subject has. Ceftaroline is effective against S.aureus germs including those that are called Methicillin Resistant Staphylococcus aureus (MRSA.)

Ceftaroline has been approved by the U.S. Food and Drug Administration (FDA) for use in adults and children with Community-Acquired Bacterial Pneumonia [a type of lung infection] and Acute Bacterial Skin and Skin Structure Infections. Ceftaroline is not yet approved for treatment in subjects with hematogenous osteomyelitis, therefore, the use of Ceftaroline in this research study is considered "investigational".

The goal of this research study is to find out what side effects there may be when children are taking Ceftaroline and to study how effective Ceftaroline is in treating bone infections due to Staphylococcus aureus in children. The investigators are also studying what the body does to the study drug, Ceftaroline, and if the doses the investigators use result in blood levels that the investigators think are going to be effective against bone infections in children. This is called pharmacokinetics (PK).

DETAILED DESCRIPTION:
This is a Phase 1/2, open-label, single-center study to determine safety and tolerability of Ceftaroline in pediatric subjects 1 to 17 years of age (inclusive) with signs and symptoms of acute hematogenous osteomyelitis at the end of intravenous therapy. After informed consent/assent is obtained, Ceftaroline will be administered intravenously. After the subject has been afebrile for at least 48 hours, has negative blood cultures, is clearly improving in general, is able to eat and drink, and is able to use or move the involved extremity, the subject may be switched to oral antibiotic administration.

The duration of subject participation from signing the informed consent form will be up to 14 months [(includes screening period (1 Day), study IV drug administration (approximately 2-14 Days), Standard of Care Oral Drug Administration (4-5 weeks) (the total maximum treatment period is typically 6 weeks), and a follow-up visit 12 months after the last dose of study drug)]. Baseline assessments for study eligibility will occur within 24 hours before the first dose of study drug. A minimum of 2 days (48 hours) of study drug administration is required.

Some of the tests and procedures completed during this study may be part of regular care for the subject's condition. Some tests and procedures will be done only for study purposes. Some regular procedures may also be completed more often as part of the research study.

Study assessments:

1. Past and Current Medical History: A detailed review of the subject's medical history, including demographics, concomitant medication review, medical/surgical history will be performed.
2. Vital Signs: Weight, height, blood pressure, pulse rate, and body temperature, will be recorded.
3. Physical Exam: Physical exam will include, evaluation of subject's overall health, examination site of infection, and assessment of subject's ability to move affected limb.
4. Safety Laboratory Assessments: Routine laboratory monitoring including liver function tests will be done 24 hours prior to enrollment and weekly during Ceftaroline treatment, and the completion of Ceftaroline treatment and at the follow-up visit. Isolate susceptibility testing will be done at baseline visit.
5. Pregnancy testing: For females of child-bearing potential, urine pregnancy will be performed prior to and after completing antibiotic treatment.
6. Pharmacokinetics Assessment: One PK blood sample will be obtained from all subjects who receive Ceftaroline fosamil.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent in writing from parent(s) or other legally acceptable representative(s) and assent from subject (if appropriate according to local requirements)
* Male or female 1 to 17 years of age, inclusive.
* Suspected hematogenous S.aureus osteomyelitis in a large bone (upper or lower extremities, pelvis) based on clinical findings and radiology results.
* One to three site(s) of osteomyelitis with expectation that transition to oral antibiotics from IV therapy will be likely prior to discharge to complete antibiotic therapy. The second or third site might be contiguous like a proximal tibia and distal femur but could also be at sites unrelated such as a distal femur and pelvic bone.
* Female subjects who have reached menarche must have a negative urine pregnancy test.
* Female subjects who have reached menarche and are sexually active must be willing to practice sexual abstinence or dual methods of birth control during treatment and for at least 28 days after the last dose of any study drug.
* Sufficient IV access to receive medication.

Exclusion Criteria:

* Received more than 24 hours of IV antibiotics prior to enrollment
* More than one bone infected
* Disseminated infection or is admitted to the pediatric intensive care unit
* Underlying condition (excludes mild eczema or reactive airways disease)
* Suspected venous thrombosis or concern for endocarditis
* Requirement for other reasons for another antibiotic potentially active against organisms commonly causing osteomyelitis in children.
* Creatinine clearance less than 50 mL/min/1.73m2 (calculated by the Schwartz formula)
* Liver transaminases greater than 3 times the upper limit of normal
* Neutropenia (less than 500 neutrophils/mm^3
* Thrombocytopenia (less than 50,000 platelets/mm^3)
* Females who are currently pregnant or breast feeding
* Hypersensitivity reaction to any Beta-lactam antibiotic
* Has had an allergic reaction to ceftaroline in the past

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2015-06-03 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon L. Kaplan, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

REFERENCES:
- See also: Physician Profile — http://www.texaschildrens.org/find-a-doctor/sheldon-l-kaplan-md

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ceftaroline Fosamil
Started | 11
Completed | 7
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Ceftaroline Fosamil
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 10.7 [2.3 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Hispanic | 6
  Race/Ethnicity: Non Hispanic | 5
  Number analyzed: Hispanic | 6
  Number analyzed: Non Hispanic | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11
Number of participants [Count of Participants; unit: Participants] | 11

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), Deaths and Discontinuations Due to Adverse Events (AEs)
Description: Evaluate the safety of Ceftaroline in pediatric subjects 1 to 17 years of age (inclusive) with acute hematogenous osteomyelitis at the end of intravenous therapy.
Time Frame: Predose and every 8 hours up to a maximum of 14 days for ceftaroline administration.
Population: One patient never received ceftaroline after enrollment because his bone biopsy showed histiocytosis.
Measure: Number; unit: incidence
Arm/Group | Ceftaroline Fosamil
Number analyzed (Participants) | 11
incidence | 1

2. Secondary Outcome: Clinical Response at the Conclusion of IV Ceftaroline
Description: Clinical response (the subject has been afebrile for at least 48 hours, has negative blood cultures, is clearly improving in general, is able to eat and drink, and is able to use or move the involved extremity) at the end of parenteral therapy (approximately days 5 to 14) by subject and by baseline pathogens although S.aureus is expected to be the predominant pathogen.
Time Frame: 2 weeks
Population: 10 patients who received ceftaroline
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftaroline Fosamil
Number analyzed (Participants) | 10
Participants | 7

3. Secondary Outcome: Clinical Outcome at the Completion of Total Therapy (IV Ceftaroline Plus Oral Antibiotics)
Description: Clinical outcome (site of infection has complete resolution of pain, swelling and warmth, normal erythrocyte sedimentation rate and C-reactive protein level and the patient is able to use the affected extremity normally and is back to normal activities) at the completion of antibiotic treatment (IV ceftaroline plus oral antibiotics).
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftaroline Fosamil
Number analyzed (Participants) | 10
Participants | 7

4. Secondary Outcome: Clinical Outcome During the One Year Follow-up Period After End of Antibiotic Treatment Which is Approximately 14 Months After Enrollment.
Description: Clinical outcome (no recurrence of pain, redness, swelling at site of original infection; absence of drainage from surgical wound; absence of pathological fracture; no other evidence of recurrence of infection at the original site of osteomyelitis and the patient is able to use the affected extremity normally and is back to normal activities) during the one year follow-up period which occurred approximately 14 month after enrollment and 12 months after completing antibiotic treatment.
Time Frame: 14 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftaroline Fosamil
Number analyzed (Participants) | 10
Participants | 7

5. Secondary Outcome: Proportion of Participants With Plasma Levels of Ceftaroline That Exceeds 1 μg/mL for Over 60% of a Dosing Interval
Description: The mean and median concentrations of ceftaroline in plasma at the end of infusion will be determined. The proportion of patients with plasma levels of Ceftaroline that exceed 1 μg/mL for over 60% of a dosing interval will be determined.
Time Frame: Blood for ceftaroline levels could be obtained once on study day 2 through day 5 post infusion of a dose of ceftaroline.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceftaroline Fosamil
Number analyzed (Participants) | 10
Participants | 10

ADVERSE EVENTS:
Time Frame: 14 months
Arm/Group | Ceftaroline Fosamil
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftaroline Fosamil (N=11)
progression of infection (Infections and infestations) | 1 (1) — 2.3 yo with MRSA osteomyelitis of left femur, tibia and septic arthritis of the hip. He received 2 doses of ceftaroline, had IR drainage of the hip but was transferred to the PICU. His blood cultures after the 2 doses of ceftaroline were negative.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/05/NCT02335905/Prot_SAP_000.pdf